CLINICAL TRIAL: NCT02130440
Title: Evaluation of the Beneficial Effects of a Nasal Spray of Resveratrol in Children With Seasonal Allergic Rhinitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Prof. Michele Miraglia del Giudice, Prof. Michele Miraglia del Giudice, University of Campania Luigi Vanvitelli
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RESV_01
Record Dates: First submitted 2014-04-25; First posted 2014-05-05 (Estimated); Last update posted 2014-05-05 (Estimated); Status verified 2014-05

CONDITIONS: Seasonal Allergic Rhinitis
Keywords: nasal obstruction; sneezing; itching; rhinorrhea; respiratory infections; wheezing
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Nasal Obstruction; Sneezing; Pruritus; Rhinorrhea; Respiratory Tract Infections; Respiratory Sounds

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Resveratrol nasal spray (Active Comparator): 2 sprays per nostril 3 times a day for a period of two months
  Interventions: Drug: Resveratrol nasal spray
- Placebo (Placebo Comparator): 2 sprays per nostril 3 times a day for a period of two months
  Interventions: Drug: Resveratrol nasal spray

INTERVENTIONS:
Drug: Resveratrol nasal spray

SUMMARY:
The aim of this study is to evaluate whether treatment with a nasal spray based on resveratrol has some benefit in patients with seasonal allergic rhinitis, mild, moderate, or severe.

DETAILED DESCRIPTION:
The aim of this study is to evaluate whether treatment with a nasal spray based on resveratrol has some benefit in patients with seasonal allergic rhinitis, mild, moderate, or severe. The primary objective is to assess whether the treatment with nasal spray based resveratrol is able to improve the allergic rhinitis symptoms during the two months of treatment. The secondary aim is to evaluate if the resveratrol nasal spray is able to reduce respiratory infections and wheezing episodes.

ELIGIBILITY:
Inclusion Criteria:

* Children of both sexes, ranging in age from 4 to 17 years
* History of seasonal allergic rhinitis, mild, moderate or severe, defined according to the ARIA guidelines in 2010, documented by recurrent episodes in the previous year and confirmed by a positive skin test results
* Written informed consent from at least one parent or a legal representative

Exclusion Criteria:

* Lack of informed consent in writing by at least one parent or a legal representative
* Concomitant disorders, such as infection of the upper (sinusitis, etc..) or lower respiratory tract, nasal surgery in the last year, abnormalities of the respiratory tract, immune diseases
* Use of antihistamines, nasal or systemic corticosteroids, leukotriene modifiers, cromolyn sodium, in the last six weeks

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2012-11; Primary Completion 2013-12 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Nasal symptom severity | two years
  Nasal symptoms (itching, sneezing, rhinorrhea, and obstruction) will be scored by a four-point scale (0=no symptom; 1=mild; 2= moderate; 3= severe) and record by parents on a daily diary card.

SECONDARY OUTCOMES:
Cough | two years
  The cough presence and severity will be assessed during the day and the night by four-point scale and recorded by parents on a daily diary card.
Wheezing | two year
  Wheezing will be assessed using the same four-point scale and record by parents on a daily diary card.
Albuterol use | two years
  The albuterol use on demand will be record by parents on a daily diary card.
Fever | two years
  The days with fever will be record by parents on a daily diary card.
School absences | two years
  School absences will be record by a diary card.
Antihistamines use | two years
  Evaluation of Cetirizine syrup on-demand use will be record by parents on a diary card
Emergency visits | two years
  Emergency room visits for respiratory problems will be record by parents on a diary card.

CONTACTS AND LOCATIONS:
Locations (1):
- Second University of Naples, Naples, Italy, Italy

REFERENCES:
- [Derived] Miraglia Del Giudice M, Maiello N, Capristo C, Alterio E, Capasso M, Perrone L, Ciprandi G. Resveratrol plus carboxymethyl-beta-glucan reduces nasal symptoms in children with pollen-induced allergic rhinitis. Curr Med Res Opin. 2014 Oct;30(10):1931-5. doi: 10.1185/03007995.2014.938731. Epub 2014 Jul 7. PMID 24983742